CLINICAL TRIAL: NCT07224711
Title: The Impact of Perioperative Lidocaine Infusions on Enhanced Recovery After Abdominal Surgery (IMPALA ERAS)
Brief Title: The Impact of Perioperative Lidocaine Infusions on Enhanced Recovery After Abdominal Surgery
Acronym: IMPALA ERAS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Danial Shams, Assistant Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 250617
Record Dates: First submitted 2025-10-21; First posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Pain; Post Operative Analgesia; Opioid Consumption, Postoperative
MeSH Terms: conditions — Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LIdocaine (Active Comparator): Participants randomized to receive 1.5 mg /kg bolus of 0.8% lidocaine Hydrochoride (HCL) in dextrose 5% in water (D5W) via IV with induction, prior to infusion started. The IV bolus will be followed by continuous IV infusion of 2 mg/minute of 0.8% lidocaine HCl in D5W intraoperatively with weight-based gradated dosing postoperatively (1-2 mg/minute)
  Interventions: Drug: Lidocaine HCl 0.8% in D5W
- Placebo (Placebo Comparator): Participants randomized to receive sodium chloride 0.9% via IV with induction, prior to infusion started. The IV bolus will be equivalent in volume to the lidocaine arm. The bolus will be followed by continuous IV infusion intraoperatively and then up to 48 hours. The continuous IV infusion will be equivalent in volume and rate to the lidocaine arm.
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Lidocaine HCl 0.8% in D5W — 1.5 mg /kg bolus of 0.8%lidocaine HCl in D5W via IV with induction, prior to infusion started. The IV bolus will be followed by continuous IV infusion of 2 mg/minute of 0.8% lidocaine HCl in D5W intraoperatively with weight-based gradated dosing postoperatively (1-2 mg/minute)
  Arms: LIdocaine
Drug: Sodium Chloride 0.9% — Sodium chloride 0.9% via IV with induction, prior to infusion started. The IV bolus will be equivalent in volume to the lidocaine arm. The bolus will be followed by continuous IV infusion intraoperatively and then up to 48 hours. The continuous IV infusion will be equivalent in volume and rate to the lidocaine arm.
  Arms: Placebo

SUMMARY:
The goal of this single-center, pragmatic, randomized, blinded, placebo-controlled trial is to evaluate the impact of intravenous (IV) lidocaine within the existing Enhanced Recovery After Surgery (ERAS)program on outcomes in patients after major abdominal surgery. The main questions the trial aims to answer are:

The primary hypothesis is that utilization of IV lidocaine as part of a perioperative multimodal pain regimen will result in a reduction in hospital Case Mix Index-Adjusted Resource Length of Stay (CARLOS).

The secondary hypotheses are that lidocaine infusion will result in a reduction in total inpatient opioid consumption (oral morphine milligram equivalents, oMMEs) and pain scores, and improved surgical outcomes (including return of bowel function, ileus, nausea, rapid responses called, surgical site infections, and ICU transfers), while also having minimal incidence of side effects (including double/blurry vision, tinnitus, sedation, and adverse events requiring early cessation).

ELIGIBILITY:
Inclusion criteria:

* Age greater than or equal to 18
* American Society of Anesthesiologists (ASA) class II-IV
* Presenting for major elective, abdominal surgery on the colorectal, emergency general surgery, urology, ventral hernia, surgical oncology, or spine services on a weekday
* First surgery in the study period (if a patient has multiple surgeries, only the first will be included)

Exclusion criteria:

* ASA class >IV
* Emergent procedures
* Allergy or any contraindication to lidocaine infusion
* Patient refusal
* Unable to receive or refusal to receive a regional nerve block
* Patients who receive an epidural due to standard of care
* Direct transfer from operating room to ICU with endotracheal tube in place
* Treating team determines patient ineligible prior to study drug administration
* Same day surgery
* Pregnancy (all women of childbearing potential are already tested as standard of care day of surgery and will be excluded from this study if found to be pregnant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2290 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Case Mix Index-Adjusted Resource Length of Stay (CARLOS) | Hospital admission to discharge (usually 4-7 days)
  The difference of CARLOS between the placebo and experimental groups in days. The Case Mix Index-Adjusted Resource Length of Stay is a hospital quality metric that standardizes average length of stay (LOS) to account for the complexity and severity of a hospital's patient population, represented by its Case Mix Index (CMI). A higher CMI indicates a more resource-intensive patient group, while a lower CMI reflects a simpler, less costly case mix.

SECONDARY OUTCOMES:
Resource Length Of Stay (RLOS) | Hospital admission to discharge (usually 4-7 days)
  Duration a patient spends in a healthcare facility as a measure of resource use
Case Mix Index | Hospital admission to discharge (usually 4-7 days)
  The difference of Case Mix Index (CMI) between the placebo and experimental groups in days. The Case Mix Index is a hospital quality metric that reflects the average clinical complexity and resource intensity of the patient population. A higher CMI indicates a more resource-intensive patient group, while a lower CMI reflects a simpler, less costly case mix.
Total consumption of inpatient opioids | Day of surgery to hospital discharge (usually 4-7 days)
  Total consumption of inpatient opioids measured in oral morphine milligram equivalents (oMME)
Pain Visual Analog Score | 0 (first pain score in Post Anesthesia Care Unit (PACU) or Intensive Care Unit(ICU)), 4, 8, 12, 24, 48, 72 hours after PACU/ICU admission and at hospital discharge
  Pain measured with an 11 point visual analog score (0 to 10) where 0 represents no pain and 10 represents the worst pain imaginable.
Incidence of surgical outcomes | Surgery to 30 days after hospital discharge
  Incidence of surgical outcomes such as bowel function, ileus, nausea, rapid response calls, surgical site infections, and Intensive Care Unit transfers
Incidence of treatment side effects | Anesthesia Induction to end of study treatment, less than or equal to 48 hours
  Incidence of treatment side effects (double/blurry vision, tinnitus, sedation and events requiring early cessation of study treatment).
Incidence of meeting early discharge milestones | hospital discharge (usually 4-7 days after surgery)
  Incidence of hospital discharge earlier than expected based on anticipated discharge day indicated at initial hospital booking

CONTACTS AND LOCATIONS:
Overall Officials: Danial Shams, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No